CLINICAL TRIAL: NCT05700032
Title: The Impact of High Mechanical Index Ultrasound Impulses on Left Ventricular Stroke Volume in Patients Receiving Intravenous Microbubbles
Brief Title: Impact of High Mechanical Index Ultrasound Impulses on Left Ventricular Stroke Volume With Intravenous Microbubbles
Acronym: MI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to clinical service demand study was withdrawn and not activated
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0134-20-FB
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- high MI (Experimental): patients receiving high MI impulses
  Interventions: Diagnostic Test: high MI impulses
- low MI (Active Comparator): patients receiving low MI impulses
  Interventions: Diagnostic Test: low MI impulses

INTERVENTIONS:
Diagnostic Test: high MI impulses — patients will receive intermittent high MI impulses(>1.0) in addition to low MI imaging. LVOT VTI will be measured at different times per protocol.
  Arms: high MI
Diagnostic Test: low MI impulses — patients will receive low MI imaging only. LVOT VTI will be measured at different times per protocol.
  Arms: low MI

SUMMARY:
This study will investigate whether applying high mechanical index (MI) impulses from a diagnostic ultrasound transducer when using ultrasound enhancing agent (UEA) microbubble infusion will result in subclinical improvement in left ventricle systolic function.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether applying high MI impulses from a diagnostic ultrasound transducer when using ultrasound enhancing agent(UEA) microbubble infusion will result in subclinical improvement in LV systolic function detected by left ventricular outflow tract velocity time integral (LVOT VTI).

ELIGIBILITY:
Inclusion Criteria:

age 19 years or older

Exclusion Criteria:

1. severe aortic valve stenosis
2. pregnant or lactating women
3. atrial fibrillation
4. very poor image quality despite contrast use.
5. unstable cardiac condition such as cardiogenic shock.
6. allergy to UEA
7. presence of right to left or bidirectional shunts.
8. Patients on mechanical circulatory support.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Left Ventricle Outflow Tract (LVOT) First Ventilatory Threshold VTI | 10 minutes
  Left Ventricle Outflow Tract (LVOT) First Ventilatory Threshold VTI

SECONDARY OUTCOMES:
stroke volume | 10 minutes
  The volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction

CONTACTS AND LOCATIONS:
Overall Officials: Swethika Harini Sundaravel, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No